CLINICAL TRIAL: NCT05739266
Title: Prediction of Pulmonary Function and Qi Deficiency Based on the Acoustic Analysis Before and After Step Test
Brief Title: Pulmonary Function and Qi Deficiency Predicted by Acoustic Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH111-REC2-036
Record Dates: First submitted 2023-02-12; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Qi-Xu; Qi Deficiency; Pulmonary Function; COPD
Keywords: Qi-Xu; Qi deficiency; Pulmonary Function; COPD; Step test; heart recovery rate
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before step test: Before step test.
  -Participants record their before-step-test voice.
- After step test: After step test.
  -Participants record their after-step-test voice.
  Interventions: Behavioral: 3 minutes step test

INTERVENTIONS:
Behavioral: 3 minutes step test — 3 minutes step test- Stair hight:20 cm, Pace: 96 steps per minute
  Groups: After step test

SUMMARY:
Acoustic analysis is a method of clinically non-invasive, low-cost, remote-operation, and can avoid direct face-to-face contact.

It has been proved by many researches in recent years that it has a high diagnostic rate in predicting diseases. Lung function is closely related to human vocalization and has the potential and need for sound analysis. From literature review, it can be inferred that the Qi deficiency constitution in TCM is related to the strength of heart and lung function.The purpose of this study is to investigate the correlation between cardiopulmonary function and Qi deficiency, and to predict the correlation between the data by computer algorithm and artificial intelligence. Furthermore, the artificial intelligence (AI) self-correction ability can be combined with sound analysis to simulate a sound analysis system that can predict cardiopulmonary function and degree of qi deficiency only through sound information.

Research motivation and questions:

1. Is the sound characteristic of an individual related to individual's qi deficiency and cardiopulmonary function?
2. Can lung function and qi deficiency be measured by sound analysis?
3. To understand the correlation between Qi deficiency and cardiopulmonary endurance index.
4. Is there any difference in sound characteristics before and after step test and does it help predicting cardiopulmonary function?

ELIGIBILITY:
Inclusion Criteria:

* Age: over 20 years old.
* Agreed and signed Informed Consent Form.

Exclusion Criteria:

* Known heart diseases, acute severe respiratory infection, severe arthritis or other orthopedic disabilities, severe hypertension, or pregnant.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Students and staffs of China Medical University, Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
FVC<80% | 10 mins
  FVC<80%
FVC>80% | 10 mins
  FVC>80%
Qi deficient | 10 mins
  Qi deficient
step test: heart rate recovery | 15 mins
  Tecumseh step test.
Voice record | 15 mins
  /a/, /e/, /i/, /o/, /u/, five seconds each, 3 times per person

CONTACTS AND LOCATIONS:
Locations (1):
- No. 2, Yude Road, North District, Taichung, Taichung City, Taiwan